CLINICAL TRIAL: NCT03578419
Title: Small-Volume Tubes to Reduce Anemia and Transfusion: A Pragmatic Stepped Wedge Cluster Randomized Trial
Brief Title: Small-Volume Tubes to Reduce Anemia and Transfusion
Acronym: STRATUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STRATUS
Record Dates: First submitted 2018-06-21; First posted 2018-07-06 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Blood Loss Anemia
Keywords: Anemia; Blood transfusion; Intensive Care Unit; Blood sampling; Stepped wedge; Red blood cells
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: A stepped wedge cluster randomized trial in which ICUs (clusters) switch from a strategy of blood collection using standard-draw tubes (control) to soft-draw tubes (intervention). In this design, the timing at which individual ICUs switch to the intervention is randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Period (Active Comparator): Standard-Volume Blood Collection Tubes
  Interventions: Device: Standard-Volume Blood Collection Tubes
- Intervention Period (Experimental): Small-Volume Blood Collection Tubes ("soft-draw")
  Interventions: Device: Small-Volume Blood Collection Tubes

INTERVENTIONS:
Device: Small-Volume Blood Collection Tubes — Small-volume vacuum (< 4 mL) ethylenediaminetetraacetic acid (EDTA), lithium-heparin, citrate, fluoride and serum blood collection tubes.
  Arms: Intervention Period
Device: Standard-Volume Blood Collection Tubes — Standard-volume (≥ 4 mL) ethylenediaminetetraacetic acid (EDTA), lithium-heparin, citrate, fluoride and serum blood collection tubes.
  Arms: Control Period

SUMMARY:
STRATUS will evaluate the use of small-volume ("soft-draw") blood collection tubes for laboratory testing in reducing anemia and transfusion in intensive care unit patients without significant adverse consequences. This is a simple, cost-neutral intervention that could improve the quality of patient care and reduce the harms of frequent laboratory testing.

DETAILED DESCRIPTION:
Blood sampling can cause significant unnecessary blood loss particularly in the intensive care unit (ICU). Blood loss contributes to anemia which is highly prevalent in the ICU and is associated with major adverse cardiovascular outcomes and death. Red blood cell (RBC) transfusions to correct anemia also have significant health risks.

Using a stepped wedge cluster randomized trial design, the specific aim of the STRATUS study is to evaluate whether the routine use of small-volume blood collection tubes reduces RBC transfusion compared to standard-volume blood collection tubes in adult ICU patients.

ELIGIBILITY:
ICUs will be eligible if they meet the following criteria:

1. Adult ICU
2. At least 14 level 2-3 ICU beds with capacity for invasive mechanical ventilation
3. Use of vacuum tubes for routine blood collection
4. Able to achieve at least 25% estimated reduction in blood volume by switching to small-volume vacuum tubes
5. Electronic administrative and health record data available for data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27411 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
RBC Transfusions | through study completion, an average of 1.5 years
  Average number of red blood cell (RBC) units transfused per patient during ICU admission among patients admitted to ICU for 48 hours or longer.

SECONDARY OUTCOMES:
Hemoglobin Concentration | through study completion, an average of 1.5 years
  Change in hemoglobin concentration from ICU admission to ICU discharge adjusted for number of RBC transfusions received
ICU and hospital length of stay | through study completion, an average of 1.5 years
  Length of stay in the ICU and hospital
ICU and hospital mortality | through study completion, an average of 1.5 years
  Mortality rates in the ICU and hospital

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Siegal, MD MSc FRCPC, Principal Investigator — Population Health Research Institute; McMaster University; Stuart Connolly, MD, Study Chair — Population Health Research Institute; McMaster University
Locations (24):
- Canada (24):
  - University of Manitoba - Health Sciences Centre, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - William Osler Health System - Brampton Civic, Brampton, Ontario
  - Joseph Brant Hospital, Burlington, Ontario
  - William Osler Health System - Etobicoke General, Etobicoke, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - London Health Sciences Centre - CCTC, London, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - St. Catharine's General Hospital, Saint Catherines, Ontario
  - Hôtel-Dieu de Lévis, Lévis, Quebec
  - CHUM - AB cardiothoracic, Montreal, Quebec
  - CHUM - CD transplants/surgical ICU, Montreal, Quebec
  - CHUM - EF neuro ICU, Montreal, Quebec
  - Maisonneuve-Rosemont, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - CHU de Quebec - Enfant-Jésus, Québec, Quebec
  - Universite de Sherbrooke - Hopital Fleurimont, Sherbrooke, Quebec
  - Universite de Sherbrooke - Hôtel-Dieu, Sherbrooke, Quebec
  - Ciuss-McQ-Chaur, Trois-Rivières, Quebec
  - CHU de Quebec - Hotel Dieu, Québec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Siegal DM, Belley-Cote EP, Lee SF, Hill S, D'Aragon F, Zarychanski R, Rochwerg B, Chasse M, Binnie A, Honarmand K, Lauzier F, Ball I, Al-Hazzani W, Archambault P, Duan E, Khwaja K, Lellouche F, Lysecki P, Marquis F, Naud JF, Shahin J, Shea J, Tsang JLY, Wang HT, Crowther M, Arnold DM, Di Sante E, Marfo G, Kovalova T, Fonguh S, Vincent J, Connolly SJ. Small-Volume Blood Collection Tubes to Reduce Transfusions in Intensive Care: The STRATUS Randomized Clinical Trial. JAMA. 2023 Nov 21;330(19):1872-1881. doi: 10.1001/jama.2023.20820. PMID 37824152